CLINICAL TRIAL: NCT01860131
Title: Evaluating Self-Management and Educational Support in Extremely Obese Patients Awaiting Multidisciplinary Bariatric Care
Brief Title: Self-Management and Educational Support in Extremely Obese Patients Awaiting Bariatric Care
Acronym: EVOLUTION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Alberta Innovates Health Solutions (Other); Alberta Health services (Other)
Responsible Party: Principal Investigator, Raj Padwal, Associate Professor of Medicine, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CIHR 201200877
Record Dates: First submitted 2013-05-17; First posted 2013-05-22 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Obesity
Keywords: bariatrics, lifestyle and behavioral modification programs
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Weight Wise Community Modules: Workshops (Active Comparator): Groups workshops (10 in total) designed to improve weight management skills and enhance self-efficacy, delivered over 3 months, prior to entering a multidisciplinary bariatric care.
  Interventions: Behavioral: Weight Wise Community Modules
- Weight Wise Community Modules: Online (Active Comparator): Online modules (13 in total) designed to improve weight management skills and enhance self-efficacy, delivered over 3 months, prior to entering a multidisciplinary bariatric care.
  Interventions: Behavioral: Weight Wise Community Modules
- Educational Written Materials (No Intervention): Educational pamphlets about healthy living and tips on self-management strategies.
  Delivered by mail 3 months prior to entering a multidisciplinary bariatric care.
  This is minimal intervention and considered the control arm.

INTERVENTIONS:
Behavioral: Weight Wise Community Modules — Program designed to educate patients regarding proper diet, exercise,and behavioural modification techniques with emphasis on increasing self-management, enhancing self-efficacy and identifying/overcoming barriers to success.
  Arms: Weight Wise Community Modules: Online; Weight Wise Community Modules: Workshops

SUMMARY:
Extreme obesity is present in 9% of the Canadian population. Extremely obese people have a high chance of developing health problems and dying early. Our national guidelines recommend that extremely obese individuals receive multidisciplinary treatment, meaning that a number of specialized care providers should be available to help administer obesity treatments to these patients.

The investigators oversee a large obesity program called the Weight Wise Obesity Program, which delivers multidisciplinary care at 5 sites in Alberta, Canada (Edmonton, Calgary, Grand Prairie, Medicine Hat, Red Deer). Wait times to enter the Weight Wise clinics range from a few months to three years depending on the site in Alberta. The investigators performed a survey of the patients on the wait list in Edmonton and discovered that they self- report extremely poor health and feel that the long wait times are partly responsible for this poor health. To try to support these patients as they wait for multidisciplinary care, the investigators designed a group based self-management intervention, consisting of Weight Wise Community Modules. Patients attend this program over three months to receive weight management education (diet, exercise, stress management, coping strategies).A web-based version of the modules is also available.

The investigators wish to determine if these modules delivered to patients prior to entering the clinic help to reduce weight, improve quality of life in the wait listed patients and also to see if going through the modules helps patients to be more ready for weight management when they reach the Weight Wise clinic. The investigators also wish to examine whether or not these modules are cost effective. If these modules are not useful, a more effective way to support wait listed patients will be sought.

DETAILED DESCRIPTION:
Background:

Extreme obesity (body mass index ≥ 35 kg/m2) affects 9% of Canadians; has tripled in prevalence in 3 decades; shortens life expectancy by 5-13 years; and is debilitating and costly. Current guidelines recommend that extremely obese patients receive treatment [consisting of intensive lifestyle modification ± bariatric (obesity) surgery] within a multidisciplinary bariatric setting. However, in Canada and other publicly funded health care settings, demand for multidisciplinary bariatric care far outstrips the capacity to provide it and so patients often face protracted, multiyear wait times. A recent study examining 150 patients on the Edmonton wait list (done at a time when the wait was several years in Edmonton) demonstrated that these patients self-report severely impaired health status (similar to those with diabetes or COPD) and strongly feel that prolonged wait times are a major contributor to their health impairments. To support these patients as they wait for more definitive management, our multidisciplinary team of clinicians, allied health professionals and decision makers have designed and implemented a Weight Wise Community Module (WWCM) program, consisting of a 3-month, 10-session group-based weight self-management intervention. In addition, a web-based version of the WWCM is now available. The WWCM program teaches self-management skills to improve diet, increase physical activity, reduce stress and increase self-efficacy - but it has not yet been evaluated. We are interested both in the outcomes after three months and after the patient has gone through the weight management clinic.The comparative clinical and cost-effectiveness of the in-person WWCM, web-based WWCM and usual care are not known.

Objectives:

To determine if an evidence-based weight-management program currently being delivered to adult (age 18 years or greater) extremely obese patients wait-listed for multidisciplinary bariatric (obesity) care in a population-based program improves clinical and humanistic outcomes, and is cost-effective.

Study Design:

This 9-month study will use a pragmatic, prospective, randomized, controlled design in which consenting extremely obese patients, newly wait listed for the Weight Wise Adult Clinic, will be randomly assigned one of three groups:

1. Weight Wise Community Modules delivered in person (9 modules delivered over 10 sessions).
2. Weight Wise Community Modules delivered on the web (13 modules, content is similar to the in-person modules)
3. Mailed Educational Pamphlets (including Canada's Guide to Health Living and tips on self-management strategies and improving readiness-to-change).

Each study arm will be comprised of 220 patients (660 total).Randomization will be performed independently of the research team by an independent organization, the EPICORE Centre.

Procedures:

Patients will be enrolled at the point of referral to each zonal program. They will have 3 months to complete the modules or review the mailed educational materials. After this, they will enter the weight management clinic in their zone. They will be followed by the study team for an additional six months while they are in the weight management clinic. Study outcomes assessments will occur at 3,6, and 9-months post randomization. If patients undergo bariatric surgery during the follow-up period, data will still be collected but they may need to be censored in the analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index (BMI) ≥ 35 kg/m2
2. Newly wait-listed for a provincial Weight Wise Adult Clinic
3. Adult age ≥ 18 years.

Exclusion Criteria:

1. Completed more than 4 Weight Wise Community Modules (web-based or group session) in previous 3 months
2. Pregnant female
3. Unable to read/write/comprehend English
4. Unable to access the web
5. Unable or unwilling to attend in-person module sessions
6. Untreated severe personality disorder, active psychosis, active substance dependence and/or major cognitive impairment
7. Participation in concurrent trial related to obesity management
8. Resides greater than 1 hour driving time to Weight Wise Clinic
9. Declined to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 651 (Actual)
Dates: Start 2013-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving 5% weight loss | 9 months
  Current consensus guidelines endorse a 5% weight loss to achieve clinically meaningful health benefits after 6-12 months of intervention.

SECONDARY OUTCOMES:
Clinical outcomes: mean 9-month change in weight | 9 months
  kg
blood pressure | 9 months
  mm hg
total cholesterol | 9 months
  mmol/L
hemoglobin A1C | 9 months
cardiovascular medications | 9 months
  number of medications
hypertension prevalence | 9 mo
diabetes prevalence | 9 mo
dyslipidemia prevalence | 9 months

OTHER OUTCOMES:
SF12 quality of life | 9 months
  total and domain scores
incremental cost-utility | 9 months
  $Cdn/QALY
Attrition rate from weight management clinic. | 9 months
EQ5D | 9 mon
  total score
WEL self efficacy scale | 9 months
  total score
readiness to change | 9 months
  visual analogue score
PHQ-8 depression scale | 9 months
  total score

CONTACTS AND LOCATIONS:
Overall Officials: Raj Padwal, MD, MSc, Principal Investigator — General Internal Medicine and Clinical Pharmacology, University of Alberta
Locations (2):
- Canada (2):
  - Alberta Health Services, Edmonton Bariatric Speciality Clinic, Royal Alexandra Hospital, Edmonton, Alberta
  - Alberta Health Services, Bariatric Specialty Clinic, Red Deer Regional Hospital, Red Deer, Alberta

REFERENCES:
- [Background] Padwal RS, Sharma AM, Fradette M, Jelinski S, Klarenbach S, Edwards A, Majumdar SR. The evaluating self-management and educational support in severely obese patients awaiting multidisciplinary bariatric care (EVOLUTION) trial: rationale and design. BMC Health Serv Res. 2013 Aug 17;13:321. doi: 10.1186/1472-6963-13-321. PMID 24059346
- [Result] Padwal RS, Klarenbach S, Sharma AM, Fradette M, Jelinski SE, Edwards A, Majumdar SR. The evaluating self-management and educational support in severely obese patients awaiting multidisciplinary bariatric care (EVOLUTION) trial: principal results. BMC Med. 2017 Mar 2;15(1):46. doi: 10.1186/s12916-017-0808-6. PMID 28249576